CLINICAL TRIAL: NCT01004341
Title: Role of Parenting Skills, Style and Family Functioning in Pediatric Weight Loss
Brief Title: Role of Parenting Skills and Parenting Style in Pediatric Weight Loss Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Brown University (Other)
Responsible Party: Principal Investigator, Kay Rhee, Assistant Professor of Pediatrics, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K23HD057299 (NIH)
Record Dates: First submitted 2009-10-20; First posted 2009-10-29 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Pediatric Obesity
Keywords: pediatric obesity; parenting style; feeding style; behavioral skills; parenting skills; family meals
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Family-based weight control (Other): Group-based family therapy for weight loss in children age 8-12 years.
  Interventions: Behavioral: Family-based behavioral weight control intervention

INTERVENTIONS:
Behavioral: Family-based behavioral weight control intervention — Standard behavioral weight control program for children ages 8-12 years old and their parents in a family-based intervention.

SUMMARY:
The purpose of this study is to evaluate the role of different parenting skills and parenting styles in the success of children enrolled in a family-based behavioral weight control program and to compare these skills and styles to those used by families with normal weight children.

DETAILED DESCRIPTION:
Pediatric overweight has nearly tripled in the past several decades and while family-based behavioral weight control programs are the mainstay of treatment, there is considerable variability in their outcomes. Parents play an important role in the success of their children, particularly by implementing new behavioral skills. However recent evidence has also suggested that parenting style, or the way a parent interacts with their child and provides emotional support and discipline, may be another key element in pediatric weight control. Our goal is to evaluate the role of specific parenting (behavioral) skills and parenting style in the success of children enrolled in a standard family-based behavioral weight control intervention. Our goal is to examine whether specific parenting (behavioral) skills and parenting style change during the intervention and whether or not this change is related to changes in the child's BMI z-score.

ELIGIBILITY:
Inclusion Criteria:

* children between and including the ages of 8-12 years old
* child BMI >= 85th percentile
* parent willing to attend all treatment meetings
* parent and child must be able to speak, read, and understand English

Exclusion Criteria:

* a family member who is participating in another weight loss program
* the child has any serious medical problem that would limit his/her participation in the study, for example, gastrointestinal diseases, cardiac disease, immune compromised state, chronic steroid use or other medication that impacts weight, developmental delays.
* child with serious food allergies that would compromise adherence to dietary recommendations
* any family member has a major psychiatric disease or organic brain syndrome
* family is going to move outside the metropolitan area within the time frame of the study

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2009-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in parenting skills and parenting style | 0 and 6 months

SECONDARY OUTCOMES:
Change in child BMI z-score | 0 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kyung E Rhee, MD, MSc, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Rhee KE, Lumeng JC, Appugliese DP, Kaciroti N, Bradley RH. Parenting styles and overweight status in first grade. Pediatrics. 2006 Jun;117(6):2047-54. doi: 10.1542/peds.2005-2259. PMID 16740847
- [Derived] Rhee KE, Jelalian E, Boutelle K, Dickstein S, Seifer R, Wing R. Warm Parenting Associated with Decreasing or Stable Child BMI during Treatment. Child Obes. 2016 Apr;12(2):94-102. doi: 10.1089/chi.2015.0127. Epub 2016 Feb 19. PMID 26895374